CLINICAL TRIAL: NCT07336589
Title: THE EFFECTS OF A COMBINED EXERCISE TRAINING AND MASSAGE THERAPY IN CHILDREN WITH FUNCTIONAL CONSTIPATION
Brief Title: COMBINED EXERCISE AND MASSAGE PROGRAM IN CHILDREN WITH FUNCTIONAL CONSTIPATION
Acronym: FC-EXMASS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Idil Sevimli (Other)
Responsible Party: Sponsor-Investigator, Zeynep Idil Sevimli, Physiotherapist, MSc (Sponsor-Investigator), Fizyofit Pilates Stüdyosu
Organization: Fizyofit Pilates Stüdyosu (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FC-EXMASS-2025
Record Dates: First submitted 2025-12-16; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Functional Constipation (FC)
Keywords: Children; Exercise Therapy; Abdominal Massage; Pelvic Floor; Non-pharmacological Treatment; Randomized Controlled Trial
MeSH Terms: interventions — Standard of Care; Educational Status; Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either an intervention group or a control group and followed in parallel throughout the study period.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants in the control group will receive standard care and education related to bowel habits and lifestyle recommendations.
  Interventions: Behavioral: Standard Care and Education
- Intervention Group (Experimental): Participants in the intervention group will receive standard care plus a combined exercise training and abdominal massage program.
  Interventions: Other: Stretching, Strengthening, and Stabilization Exercises; Other: Abdominal Massage (I Love You Technique); Behavioral: Standard Care and Education; Other: Pelvic Floor Muscle Training; Other: Breathing Exercises

INTERVENTIONS:
Other: Stretching, Strengthening, and Stabilization Exercises — Children will complete exercises to improve flexibility, muscle strength, and trunk stability.
  Arms: Intervention Group
Other: Abdominal Massage (I Love You Technique) — Gentle abdominal massage will be applied following the colon pathway to support bowel movement.
  Arms: Intervention Group
Behavioral: Standard Care and Education — Children and their parents will receive education about bowel function and lifestyle guidance on diet, fluid intake, toileting habits, and physical activity.
Other: Pelvic Floor Muscle Training — Children will practice fast and slow pelvic floor contractions to improve muscle strength and endurance.
  Arms: Intervention Group
Other: Breathing Exercises — Children will perform simple diaphragmatic breathing exercises daily to support abdominal and pelvic muscle coordination.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to learn if a combined exercise and abdominal massage program improves bowel function and daily well-being in children with functional constipation. Researchers will compare this program with standard care by measuring bowel symptoms, rectal size, pelvic floor strength, trunk endurance, and quality of life.

DETAILED DESCRIPTION:
This clinical trial includes children with functional constipation. Participants will be randomly assigned to either a combined exercise and abdominal massage program or to standard care and education.

Children in the program group will take part in guided exercise sessions and receive abdominal massage, while the standard care group will receive routine follow-up and advice on bowel habits.

Researchers will measure bowel symptoms, bowel movement patterns, rectal diameter, pelvic floor muscle function, trunk muscle endurance, and quality of life before and after the program.

The results may help improve safe, non-drug treatment options for children with constipation.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-18 years
* Diagnosed with functional constipation according to Rome IV criteria
* Voluntary participation with written informed consent obtained from parents or legal guardians

Exclusion Criteria:

* Refusal to participate
* Presence of congenital conditions (e.g., Down syndrome, Hirschsprung disease)
* Endocrine or metabolic disorders (e.g., hypothyroidism, diabetes mellitus, diabetes insipidus)
* Neurological or psychiatric disorders (e.g., spina bifida, cerebral palsy, autism spectrum disorders)
* History of abdominal surgery within the last year
* Presence of herniation or open wounds in the abdominal massage area

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rectal Diameter (measured by ultrasound) | Baseline and after eight weeks
  Rectal diameter will be measured using abdominal ultrasonography to assess rectal distension related to functional constipation. Measurements will be performed before the intervention and at the end of the eight-week program. Changes in rectal diameter will be used to evaluate the effectiveness of the combined exercise and abdominal massage program.
Constipation Symptoms (Rome IV Diagnostic Criteria) | Baseline and after eight weeks
  Constipation symptoms will be assessed using the Rome IV diagnostic criteria for functional constipation, including bowel movement frequency, fecal incontinence, painful or difficult defecation, stool withholding behavior, and presence of large stools.

SECONDARY OUTCOMES:
Bowel Function (Bowel Diary + Bristol Stool Scale) | Baseline and after eight weeks
  Bowel function will be evaluated using a 7-day bowel diary including stool frequency and stool consistency (Bristol Stool Scale, Types 1-7). The diary will be completed for one week at baseline and for one week after the 8-week program.
Pelvic Floor Function | Baseline and after eight weeks
  Pelvic floor muscle function will be evaluated using the Oxford Scale adapted for children. Muscle contraction strength will be graded during a clinical assessment.
Quality of Life (Visual Analog Scale) | Baseline and after eight weeks
  Children's and parents' quality of life will be measured using a Visual Analog Scale ranging from zero to ten, with higher scores indicating greater impact of constipation on daily life.
Perceived Improvement (9-Point Patient Global Impression of Change Scale) | After eight weeks
  Perceived improvement will be evaluated using the 9-point Patient Global Impression of Change Scale. Parents will rate their child's overall change in constipation symptoms compared to the start of the study, with higher scores indicating greater improvement.
Treatment Adherence (Visual Analog Scale) | After eight weeks
  Adherence to treatment recommendations will be evaluated using a Visual Analog Scale completed by parents, with higher scores indicating better adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep I sevimli, PT, MSc, Principal Investigator — Fizyofit Pilates Stüdyosu / Ankara Bilkent City Hospital
Locations (1):
- Ankara Bilkent City Hospital - Pediatric Surgery Clinic, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No